CLINICAL TRIAL: NCT01494051
Title: Fatty Acid Oxidation and Body Weight Regulation in Long-chain Fatty Acid Oxidation Disorders.
Brief Title: High Protein Diet in Patients With Long-chain Fatty Acid Oxidation Disorders
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Melanie B Gillingham, Assistant Professor, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DK71869-2
Record Dates: First submitted 2011-12-14; First posted 2011-12-16 (Estimated); Results first posted 2020-04-21 (Actual); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Very Long-chain Acyl-CoA Dehydrogenase Deficiency; Trifunctional Protein Deficiency; Carnitine Palmitoyltransferase 2 Deficiency; Long-chain 3-hydroxyacyl-CoA Dehydrogenase Deficiency
Keywords: fatty acid oxidation disorders
MeSH Terms: conditions — VLCAD deficiency; Trifunctional Protein Deficiency With Myopathy And Neuropathy; Carnitine palmitoyl transferase 2 deficiency | interventions — Diet, Fat-Restricted; Diet, High-Protein Low-Carbohydrate; Diet, High-Protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High carbohydrate diet (Active Comparator): Diet composition of 10% long-chain fatty acids, 20% medium-chain triglycerides, 12% protein and 68% carbohydrate is the current standard of care in long-chain fatty acid oxidation disorders.
  Interventions: Behavioral: Diet counseling
- High protein diet (Experimental): Diet composition of 10% long-chain fatty acids, 20% medium chain triglycerides, 25% protein and 45% carbohydrate is the comparison diet. Fat content is the same between treatments; only the carbohydrate to protein ratio varies.
  Interventions: Behavioral: Diet counseling

INTERVENTIONS:
Behavioral: Diet counseling — Subjects counseled how to follow either the high carbohydrate diet or the high protein diet for 4 months at home.
  Other Names: low fat diet; high carbohydrate diet; high protein diet

SUMMARY:
The study also determines if eating a diet higher in protein alters body composition, energy balance and metabolic control among patients with a long-chain fatty acid oxidation disorder.

DETAILED DESCRIPTION:
At baseline, the amount of muscle and fat in the whole body and inside the liver and muscle will be measured. All subjects will complete a moderate treadmill exercise test and a test to determine how they use sugar (oral glucose tolerance test). The amount and type of energy burned by each subject will be measured. Subjects will be randomly assigned to follow either a high carbohydrate diet or a reduced carbohydrate, high protein diet for 4 months. At the end of 4 months, the tests will be repeated.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of a long-chain fatty acid oxidation disorder including VLCAD, CPT2, LCHAD or TFP deficiency
* 7 years old or greater
* able to comply with diet guidelines

Exclusion Criteria:

* pregnant
* enrolled in another study that alters diet composition
* cannot complete treadmill exercise study

Ages: 7 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2006-01; Primary Completion 2009-09 (Actual); Study Completion 2010-01 (Actual)

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | High Carbohydrate Diet | High Protein Diet
Started | 6 | 7
Completed | 6 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Carbohydrate Diet | High Protein Diet | Total
Number analyzed (Participants) | 6 | 7 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 14 (5) | 17 (10) | 16 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 4 | 3 | 7
Region of Enrollment [Number; unit: participants]
  North America | 6 | 6 | 12
  Sweden | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Energy Expenditure
Description: does energy expenditure and substrate oxidation differ between subjects randomized to the high carbohydrate versus the high protein diet? We measured resting energy expenditure with indirect calorimetry and estimated substrate oxidation with indirect calorimetry results and urine urea nitrogen excretion. We also measured total energy expenditure with doubly labeled water.
Time Frame: change from baseline after 4 months of treatment
Measure: Mean (Standard Deviation); unit: kcal
Arm/Group | High Carbohydrate Diet | High Protein Diet
Number analyzed (Participants) | 6 | 7
kcal | 2045 (273) | 2343 (507)

2. Secondary Outcome: Body Composition
Description: does body composition change more among subjects randomized to the high protein diet compared to the high carbohydrate diet? We measured body composition at baseline and again at the end of the study by DEXA - dual energy x-ray absorptiometry.
Time Frame: change from baseline to 4 months of treatment
Measure: Mean (Standard Deviation); unit: change in kg
Arm/Group | High Carbohydrate Diet | High Protein Diet
Number analyzed (Participants) | 6 | 7
change in kg
  Lean Mass | -0.75 (1.34) | 0.78 (1.17)
  Fat Mass | 0.51 (4.34) | 0.43 (0.9)

ADVERSE EVENTS:
Arm/Group | High Carbohydrate Diet | High Protein Diet
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/7
Other Adverse Events (participants affected / at risk) | 0/6 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No